CLINICAL TRIAL: NCT01042847
Title: The Effect of Genetic Polymorphisms in Indoleamine 2, 3-Dioxygenase in Epithelial Ovarian Cancer
Brief Title: How Our Immune System Can Help Fight Cancer
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Jeannine Villella DO, Prinicipal Investigator, Winthrop University Hospital
Other Study IDs: 09316
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Cancer
Keywords: ovarian
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — surgical tissue ascites fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
There is growing evidence that our immune system can help fight cancer. This has stimulated interest in the development and application of tumor vaccines for several human solid tumors, including epithelial ovarian cancer (EOC). A major obstacle to the development of these vaccines is that there are specialty cells called regulatory T cells that prevent the immune system from attacking all of our organs. These regulatory T cells also prevent our immune system for attacking cancer cells.

Indoleamine 2,3-dioxygenase (IDO), an enzyme that degrades an essential amino acid tryptophan that is necessary for T cells to multiply, however regulatory T cells are less susceptible to low levels of tryptophan, and can still multiply. This allows cancer growth and progression. This may be explained by genetic polymorphisms (changes) in the IDO gene, which may alter its function. Five of these changes in the IDO gene have been described. In this research project, we are asking if you would donate a small piece of your tumor and ascites to see if we can examine your IDO gene in the tumor cells and see if any of these gene changes are present. We hope that this will help us understand how the immune system works in EOC.

We hypothesize that genetic polymorphisms within the IDO gene alter its enzymatic activity and affect the outcome of ovarian cancer patients. These findings have the potential to translate into a method for predicting successful immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* females aged 20-90 who are having surgery to confirm epithelial ovarian cancer.

Exclusion Criteria:

* patients who have a diagnosis of non-epithelial histology.

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed epithelial ovarian cancer (EOC) who have had surgical resection for their disease will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2010-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To examine the association of indoleamine 2,3-dioxygenase (IDO) genetic polymorphisms with clinical outcomes of ovarian cancer. | one year

SECONDARY OUTCOMES:
To correlate IDO activity with gene polymorphisms by measuring tryptophan/kynurenine ratios in the ascites of epithelial ovarian cancer patients. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine A Villella, D.O., Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States